CLINICAL TRIAL: NCT05274932
Title: Neuromuscular Responses, Pain Intensity and Perceived Exertion of Resistance Exercise With Blood Flow Restriction in Patients With Severe Knee Osteoarthritis
Brief Title: Exercise With Blood Flow Restriction in Knee Osteoarthritis
Acronym: BFROA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, José Casaña Granell, Head of the Physiotherapy Department, University of Valencia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OA-22-01
Record Dates: First submitted 2022-02-15; First posted 2022-03-11 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Electromyography; Muscle Activity; Resistance Training
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Active Comparator): Knee extensions with 30% 1RM and no occlusion pressure.
  Interventions: Other: BFR resistance exercise
- BFR at 40% AOP (Experimental): Knee extensions with 30% 1RM and BFR at 40% AOP.
  Interventions: Other: BFR resistance exercise
- BFR at 80% AOP (Experimental): Knee extensions with 30% 1RM and BFR at 80% AOP.
  Interventions: Other: BFR resistance exercise

INTERVENTIONS:
Other: BFR resistance exercise — 4 sets (30, 15, 15, 15 reps).

SUMMARY:
The purpose of this study is to evaluate the neuromuscular responses, pain intensity and rate of perceived exertion in patients with severe knee osteoarthritis in a preoperative setting with low-load resistance training with blood flow restriction at different levels of arterial occlusion pressure.

ELIGIBILITY:
Inclusion Criteria:

* men and women above 55 years old.
* diagnosed with severe knee osteoarthritis.
* scheduled for unilateral TKA surgery in a local hospital during 2021- 2022.

Exclusion Criteria:

* pain in the contralateral limb (maximum pain, ≥80 of 100 mm on a VAS during daily activities).
* another hip or knee joint replacement in the previous year.
* any medical condition in which exercise was contraindicated.
* participated in exercise programs (>2 days/week, training at intensities of 10-15RM) in the 6 months prior to the study.
* history of stroke, brain surgery, major depression, or any self-perceived cognitive alterations that could affect the performance of dual tasks.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Self-reported pain intensity (Visual Analogue Scale (VAS) Scale 0-10) | Pre exercise, immediate post set, immediate post session, and 10 minutes after session.
  Change from baseline to the end of the session, and the change between the treatment group and the placebo group.
Pressure pain thresholds | Pre exercise, immediate post session, and 10 minutes after session.
  Change from baseline to the end of the session, and the change between the treatment group and the placebo group.
HDsEMG | During each experimental session and during each exercise condition.
  Change between baseline and exercise, and the change between the treatment group and the placebo group.

SECONDARY OUTCOMES:
Tampa Scale of Kinesiophobia (TSK 11) | Pre session.
  Its score range is 11-44, with higher scores reflecting worse condition.
Pain Catastrophizing Scale (PCS) | Pre session.
  People are asked to indicate the degree to which they have certain thoughts and feelings when they are experiencing pain using the 0 (not at all) to 4 (all the time) scale. A total score is yielded (ranging from 0-52), along with three subscale scores assessing rumination, magnification and helplessness, with higher scores reflecting worse condition.
Chronic Pain Self-Efficacy Scale (CPSS) | Pre session.
  The Chronic Pain Self-Efficacy Scale (CPSS) is designed to measure chronic pain patients' perceived self-efficacy to cope with the consequences of chronic pain. The CPSS measures three domains of pain self-efficacy: pain management, physical functioning, and coping with symptoms. A total score is yielded (ranging from 220-2200), with higher scores reflecting a better condition.
WOMAC questionaire for patients with hip or knee osteoarthritis. | Pre session.
  The WOMAC is a disease-specific self-administered questionnaire for patients with hip or knee osteoarthritis. It has a multidimensional scale made up of 24 items grouped into three dimensions: pain (5 items), stiffness (2 items) and physical function (17 items). For each item, it uses a Likert scale with five response levels, representing different degrees of intensity (none, mild, moderate, severe or extreme) that are scored from 0 to 4. The final score for the WOMAC is determined by adding the aggregate scores for pain, stiffness and function. The higher the score, the worse the patient's condition.
Heart Rate | Pre exercise, immediate post set, immediate post session, and 10 minutes after session.
  Change from baseline to the end of the session, and the change between the treatment group and the placebo group.
Rating of perceived exertion (RPE) based on Borg's CR10 scale | Immediate post exercise.
  The Borg CR10 scale is a tool for measuring an individual's effort and exertion during physical work. It is a very simple numerical list from 0 (no exertion at all) to 10 (maximal intensity of activity). Participants are asked to rate their exertion on the scale during the activity, combining all sensations and feelings of physical stress and fatigue. They are told to disregard any one factor such as leg pain or shortness of breath but to try to focus on the whole feeling of exertion.

CONTACTS AND LOCATIONS:
Overall Officials: José Casaña, Principal Investigator — University of Valencia; Joaquín Calatayud, Study Chair — University of Valencia
Locations (1):
- Clinic Universitary Hospital of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ogrezeanu DC, Lopez-Bueno L, Sanchis-Sanchez E, Carrasco JJ, Cuenca-Martinez F, Suso-Marti L, Lopez-Bueno R, Cruz-Montecinos C, Martinez-Valdes E, Casana J, Calatayud J. Neuromuscular Responses and Perceptions of Health Status and Pain-Related Constructs in End-Stage Knee Osteoarthritis During Resistance Training With Blood Flow Restriction. J Strength Cond Res. 2024 Apr 1;38(4):762-772. doi: 10.1519/JSC.0000000000004680. Epub 2023 Dec 13. PMID 38090743